CLINICAL TRIAL: NCT02584127
Title: Tobacco-Related Disease Prevention Among Korean Americans
Acronym: CFCHKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Joel Moskowitz, Director, Center for Family and Community Health, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CFCHKA
Record Dates: First submitted 2015-10-20; First posted 2015-10-22 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Smoking Cessation
Keywords: Smoking; cessation; Internet program
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High reinforcement cessation program (Experimental): The High Reinforcement (HR) condition included five monthly, online interim surveys with financial incentives for these assessments and also for program completion. All participants completed an eligibility survey and a baseline survey. All participants were offered a financial incentive to complete the six-monh followup survey. All participants were provided access to a six step, cognitive-behavioral smoking cessation program self-administered online.
  Interventions: Behavioral: high reinforcement cessation program
- Low reinforcement cessation program (Experimental): Participants in the Low Reinforcement (LR) condition participants completed an eligibility survey and a baseline survey. All participants were offered a financial incentive to complete the six-monh followup survey. All participants were provided access to a six step, cognitive-behavioral smoking cessation program self-administered online.
  Interventions: Behavioral: low reinforcement cessation program

INTERVENTIONS:
Behavioral: high reinforcement cessation program — Six-step, self-administered, internet smoking cessation program with high reinforcement.
  Arms: High reinforcement cessation program
Behavioral: low reinforcement cessation program — Six-step, self-administered, internet smoking cessation program with low reinforcement.
  Arms: Low reinforcement cessation program

SUMMARY:
The study evaluates the effectiveness of an internet-based smoking cessation program for Korean Americans.

DETAILED DESCRIPTION:
Smoking is prevalent among Korean American men. Quitting is Winning, an internet-based, cognitive-behavioral smoking cessation program, was developed using community-based participatory research principles.

A randomized controlled trial was used to evaluate whether participants were more likely to complete the program and quit smoking at 6-month follow-up with additional reinforcement including financial incentives for program completion and interim surveys.

ELIGIBILITY:
Inclusion Criteria:

* self-identified Korean American ethnicity
* age 18 years or older
* daily smoker (i.e., smoked at least one cigarette per day during the previous seven days)
* current U.S. resident
* valid email address
* regular internet access.

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2009-09; Primary Completion 2013-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
smoking status | six month followup
  self-reported smoking status at 6-month followup

SECONDARY OUTCOMES:
program completion | six months
  Percentage of participants who completed the online smoking cessation program

CONTACTS AND LOCATIONS:
Locations (1):
- Joel Moskowitz, Berkeley, California, United States

REFERENCES:
- [Derived] Moskowitz JM, McDonnell DD, Kazinets G, Lee HJ. Online smoking cessation program for Korean Americans: Randomized trial to test effects of incentives for program completion and interim surveys. Prev Med. 2016 May;86:70-6. doi: 10.1016/j.ypmed.2016.01.019. Epub 2016 Feb 1. PMID 26845375